CLINICAL TRIAL: NCT07174674
Title: Saturation and Nursing Interventions in Patients Receiving Supplemental Oxygen Therapy During the First Night After Metabolic and Bariatric Surgery
Brief Title: Desaturations and Nursing Interventions in Patients Receiving Supplemental Oxygen Therapy After Metabolic and Bariatric Surgery
Acronym: SATBAR
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-2107
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea (OSA); Bariatric Surgery
Keywords: obstructive sleep apnea; bariatric surgery; oxygen therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All study participants: Alle study participants will receive standard of care.

SUMMARY:
The goal of this observational study is to learn about the effect of supplemental oxygen therapy during the first night after bariatric and metabolic surgery in a population that is not (routinely) tested for obstructive sleep apnea preoperatively.

The main question to answer in this study is:

How many desaturations occur while participants receive supplemental oxygen therapy and how many, and what type of nursing interventions are needed? Another question we want to answer is: are there characteristics that seems to increase the risk of developing a desaturation?

DETAILED DESCRIPTION:
This is a prospective observational study that aims to characterize the number of desaturations and nursing interventions in a population with a unknown structive sleep apnea status receiving supplemental oxygen therapy during the first night after metabolic and bariatric surgery. The secondary aim is to to identify patient characteristics that are associated with a higher risk of developing desaturations.

Methods:

Participants receive standard of care, which includes 2 liters of supplemental oxygen therapy during the first postoperative night after metabolic and bariatric surgery while being continously monitored.

The desaturations, saturation and number and type of nursing intervention were collected along with patient characteristics (see outcomes) Sample size: A population proportion sample size was used, a CI 95%, margin of error 5% , proportion of 0.50, gave a required sample size of 385 participants.

Mann Whitney U-test (continuous data) and Fishers exact test (categorical data) are used to compare spo2 and nursing interventions between participants with and without desaturations.

Binary logistic regression will be used to estimate the risk for developing desaturations.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing primary metabolic and bariatric surgery
* Overnight hospital stay

Exclusion Criteria:

* Undergoing secundary metabolic and bariatric surgery (e.g. redo surgery)
* Having treated obstructive sleep apnea (CPAP, oral application)
* Having chronic obstructive pulmonary disease
* No overnight hospital stay at the nursing ward (same-day discharge or overnight stay at medium or intensive care)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary bariatric and metabolic surgery, with a overnight stay at the nursing ward of Rijnstate Hospital (Arnhem, the Netherlands). With exclusion of patients with treated OSA or diagnosis of chronic obstructive pulmonary disease.
Sampling Method: Probability Sample
Enrollment: 563 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

PRIMARY OUTCOMES:
Number of desaturations per patient | First postoperative night
  Participants were continuously monitored and all desaturations (spo2<90%) were collected.
Number of nursing interventions | First postoperative night
  If nurses had to intervene because of a desaturation or to prevent a desaturation (e.g. waking patient, putting back nasal cannula, increasing oxygen flow)
Type of nursing intervention | First postoperative night
  which nursing intervention the nursed provided was documented on a form (e.g. putting back nasal cannula, increasing oxygen flow, jaw thrust)

SECONDARY OUTCOMES:
The effect of the patient characterisic "sex" on the risk of developing desaturations | First postoperative night
The effect of the patient characterisic "age" on the risk of developing desaturations | First postoperative night
  Age on day of surgery
The effect of the patient characterisic "body mass index" on the risk of developing desaturations | First postoperative night
  Body mass index on day of surgery
The effect of the patient characterisic "smoking status" on the risk of developing desaturations | First postoperative night
  Somking status before surgery
The effect of the patient characterisic "chronic benzodiazepine use" on the risk of developing desaturations | First postoperative night
  Use of benzodiazepine at home
The effect of the patient characterisic "diabetes mellitus type 2" on the risk of developing desaturations | First postoperative night
  Preoperative diabetes mellitus type 2 status (yes/no)
The effect of the patient characterisic "hypertension" on the risk of developing desaturations | First postoperative night
  Preoperative hypertension status (yes/no)
The effect of the patient characterisic "dyslipidemia" on the risk of developing desaturations | First postoperative night
  Preoperative dyslipidemia status (yes/no)
The effect of operating time on the risk of developing desaturations | First postoperative night
  Duration of the surgery
The effect postoperatively used morphine milligram equivalent on the risk of developing desaturations | First postoperative night
  The postoperative used opioid were converted to oral morphine milligram equivalent
The effect intraoperatively used morphine milligram equivalent on the risk of developing desaturations | First postoperative night
  The intraoperative used opioid were converted to oral morphine milligram equivalent
The effect of rocuronium on the risk of developing desaturations | First postoperative night
  The intraoperative used dose of rocuronium
The effect of sugammadex on the risk of developing desaturations | First postoperative night
  The intraoperative use of sugammadex

OTHER OUTCOMES:
Saturation during the night | First postoperative night
  Every 10 minutes a mean saturation from the continuous monitoring was was saved.

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Hazebroek, MD, PhD, Principal Investigator — Vitalys obesity clinic, part of Rijnstate Hospital
Locations (1):
- Vitalys obesity clinic, part of Rijnstate Hospital, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Sharing of IPD is not necessary